CLINICAL TRIAL: NCT04376593
Title: 18F-αvβ6-binding-peptide PET/CT in Patients Post SARS CoV2 Infection
Brief Title: PET/CT Imaging in COVID-19 Patients
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1592298
Record Dates: First submitted 2020-05-03; First posted 2020-05-06 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: COVID-19; SARS-CoV-2 Infection
Keywords: COVID-19; SARS-CoV2 infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-αvβ6-BP (Experimental): Following a 10 mCi (±20%) intravenous injection (IV) of 18F-αvβ6-BP, PET/CT images will be acquired at 60 minutes. Baseline blood samples will be drawn and banked. Vital sign (VS) measurements (heart rate, respiratory rate, blood pressure and temperature) monitored throughout. Region-of-interest analysis (ROI) will be performed in the lung. Each participant will undergo up to 3 18F- αvβ6-BP PET/CT scans over a 6-month timeframe.
  Interventions: Drug: 18F-αvβ6-BP

INTERVENTIONS:
Drug: 18F-αvβ6-BP — Subjects will be injected once per imaging session (a maximum of 3 imaging sessions) with up to 10 mCi (±20%) of 18F-αvβ6-BP as a rapid intravenous bolus (within 30 secs).

SUMMARY:
This is a PET/CT study using the 18F-αvβ6-binding-peptide.The goal of this study is to evaluate this peptide in patients after infection with SARS CoV2.

DETAILED DESCRIPTION:
The goal of the study is to to acquire 18F-αvβ6-BP PET/CT images in patients diagnosed with SARS CoV2 and to demonstrate the ability of 18F-αvβ6-BP to detect lung damage.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age ≥ 18 yrs
* Diagnosed with SARS CoV2
* Must have 2 sequential COVID negative tests prior to each scan
* Must have no previous lung disease prior to SARS CoV2 infection
* Lung image (Xray or CT) taken during infectious/ diagnosis period
* Will sign the IRB-approved consent form
* Able to remain motionless for up to 30-60 minutes per scan.

Exclusion Criteria:

* Life expectancy <3 mo
* Women who are pregnant or breast-feeding
* Patients who cannot undergo PET/CT scanning because of weight limits(>350lbs)
* Lack of availability for follow-up assessments
* Re-infection with SARS CoV2 between scan sessions
* Other active infectious respiratory illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Administration of 18F-αvβ6-BP | baseline
  Completion of administration of 18F-αvβ6-BP in SARC CoV2 patients
Administration of 18F-αvβ6-BP | 3 months
  Completion of administration of 18F-αvβ6-BP in SARC CoV2 patients
Administration of 18F-αvβ6-BP | 6 months
  Completion of administration of 18F-αvβ6-BP in SARC CoV2 patients

SECONDARY OUTCOMES:
Determine whether 18F-αvβ6-BP demonstrates accumulation in lung damage | baseline
  Uptake of 18F-αvβ6-BP in lung damage will be measured by PET
Determine whether 18F-αvβ6-BP demonstrates accumulation in lung damage | 3 months
  Uptake of 18F-αvβ6-BP in lung damage will be measured by PET
Determine whether 18F-αvβ6-BP demonstrates accumulation in lung damage | 6 months
  Uptake of 18F-αvβ6-BP in lung damage will be measured by PET

OTHER OUTCOMES:
Determine whether 18F-αvβ6-BP accumulation in lung correlates to lung damage as indicated on CT. | baseline
  Uptake of 18F-αvβ6-BP in lung measured by PET will be compared to lung damage as indicated on CT.
Determine whether 18F-αvβ6-BP accumulation in lung correlates to lung damage as indicated on CT. | 3 months
  Uptake of 18F-αvβ6-BP in lung measured by PET will be compared to lung damage as indicated on CT.
Determine whether 18F-αvβ6-BP accumulation in lung correlates to lung damage as indicated on CT. | 6 months
  Uptake of 18F-αvβ6-BP in lung measured by PET will be compared to lung damage as indicated on CT.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-study-of-the-experimental-petct-radiotracer-18f-avb6-binding-peptide-after-covid-19-coronavirus-infection-935076/